CLINICAL TRIAL: NCT01599767
Title: Spaulding-Harvard Spinal Cord Injury (SH-SCI) Study: Effects of tDCS on Chronic Pain in Spinal Cord Injury.
Brief Title: Spaulding-Harvard Model System: Effects of Transcranial Direct Current Stimulation (tDCS) on Chronic Pain in Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Principal Investigator, Felipe Fregni, Associate Professor, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011-p-002353
Record Dates: First submitted 2012-02-08; First posted 2012-05-16 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Spinal Cord Injury; Chronic Pain; Neuropathic Pain
Keywords: transcranial stimulation; direct current
MeSH Terms: conditions — Spinal Cord Injuries; Chronic Pain; Neuralgia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (Experimental): Subjects will undergo 20 minutes active tDCS.
  Interventions: Device: Transcranial direct current stimulation (tDCS)
- Sham tDCS (Sham Comparator): Subjects will undergo 20 minutes of sham stimulation.
  Interventions: Device: Transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS) — Subjects will undergo 15 sessions of tDCS stimulation (either active or sham), 1x per day at 20 minutes per session.
  Other Names: 1x1 low-intensity direct current stimulator; Soterix Medical

SUMMARY:
The purpose of this study is to see the effects of transcranial direct current stimulation (tDCS) on the pain associated with spinal cord injury. This study is part of the Spaulding-Harvard Model System. The investigators hypothesize that there will be a decrease in pain levels with active stimulation, when compared to sham stimulation, using a 3 week stimulation schedule- 1 week of stimulation (5 consecutive days) followed by 2 weeks of stimulation (10 consecutive days) after a 3-month follow up visit. The subject will also have follow ups at 2, 4 and 8 weeks after the second course of stimulation.

If a subject receives sham during the experiment, he/she may enroll in an open-label portion of the study and receive 10 days of active stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* History of moderate to severe sublesional pain

Exclusion Criteria:

* Active alcohol or drug dependence, as self-reported
* A history of bipolar disorder or psychosis, as self-reported
* Inability to travel to the study site,
* Current use of any of the following anti-epileptic medications or dopaminergic medications known to reduce or inhibit the benefits of tDCS treatment [53]: carbamazepine, oxcarbazepine, phenytoin, ropinirole (Requip), pramipexole (Mirapex), and cabergoline (Dostinex),
* The following contradictions to tDCS: implanted metal plates in the head, or deep brain stimulator (spinal cord implants, including baclofen pumps, are not a contraindication as cranial currents do not reach the spinal cord [24]).
* Pregnancy at time of enrollment
* Current use of ventilator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2011-12; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in Pain Scale | Measured for approximately 6 months
  Determine whether anodal transcranial direct current stimulation is effective in reducing pain in subjects with chronic sublesional neuropathic pain due to spinal cord injury, as measured by changes in the Brief Pain Inventory (BPI) from baseline to follow-up (up to 2 months after the final stimulation session).

SECONDARY OUTCOMES:
Changes in Quality of Life Scale | Measured for approximately 6 months
  Determine whether anodal transcranial direct current stimulation is effective in increasing quality of life in subjects with chronic neuropathic sublesional pain due to spinal cord injury, as measured by changes in the Satisfaction with Life Scale (SWLS), from baseline to follow-up (up to 2 months after the final stimulation session).
Changes in Mood Scale | Measured for approximately 6 months
  Determine whether anodal transcranial direct current stimulation is effective in improving mood in subjects with chronic neuropathic sublesional pain due to spinal cord injury, as measured by changes in the Patient Health Questionnaire-9 (PHQ9), from baseline to follow-up (up to 2 months after the final stimulation session).

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Fregni, MD PHD MPH, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Thibaut A, Carvalho S, Morse LR, Zafonte R, Fregni F. Delayed pain decrease following M1 tDCS in spinal cord injury: A randomized controlled clinical trial. Neurosci Lett. 2017 Sep 29;658:19-26. doi: 10.1016/j.neulet.2017.08.024. Epub 2017 Aug 16. PMID 28822837
- See also: Spaulding-Harvard SCI Model System Website — http://www.sh-sci.org